CLINICAL TRIAL: NCT06970665
Title: A Phase 3/4, Multicenter, Single-arm Clinical Study to Assess the Safety of Intravitreal Administration of ASP3021 in Participants in Japan With Geographic Atrophy Secondary to Age-related Macular Degeneration
Brief Title: A Study About the Safety of ASP3021 Eye Injections and if They Help People in Japan With Vision Loss From Age-related Macular Degeneration
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3021-CL-3001; jRCT2031250086 (Registry Identifier: jRCT)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Geographic Atrophy; Age-Related Macular Degeneration
Keywords: avacincaptad pegol; IZERVAY; ASP3021
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ASP3021 (Experimental): Participants in Japan with Geographic Atrophy (GA) secondary to Age-related Macular Degeneration
  Interventions: Drug: avacincaptad pegol

INTERVENTIONS:
Drug: avacincaptad pegol — intravitreal injection
  Other Names: ASP3021; IZERVAY

SUMMARY:
Age-related macular degeneration (AMD) is an eye disease which causes people to lose their vision over time. AMD damages the macula, which is in the middle of the retina - the light sensitive part at the back of the eye. In AMD, the cells in the macula die over time, usually over several years, leading to vision loss. When AMD gets worse, it can turn into either geographic atrophy (GA), neovascular AMD, or both.

This study is for people in Japan of 40 years of age or older, who have geographic atrophy.

The main aim of this study is to collect information about the safety of ASP3021 and how well people tolerate treatment with ASP3021.

During the study, people will receive monthly injections of ASP3021 for 12 months. ASP3021 is given by injection into the affected eye. This procedure is called an intravitreal injection.

People will be in the study for about 1 year. People will visit their study clinic several times for health checks.

DETAILED DESCRIPTION:
IZERVAY has received marketing approval in Japan. The study will continue as a post marketing study in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participant has non-foveal central point involvement geographic atrophy (GA) secondary to age-related macular degeneration (AMD).
* Participant has total GA area ≥ 2.0 and ≤ 17.5 mm^2 (1 and 7 disc areas [DA] respectively), determined by fundus autofluorescence (FAF) screening images.
* If participant has multifocal GA, at least one focal lesion should measure ≥ 1.25 mm^2 (0.5 DA).
* Participant has GA in part within 1500 microns from the fovea center point.
* Participant has GA that must be able to be photographed in its entirety.
* Participant has best corrected visual acuity (BCVA) between 20/25 and 20/320, inclusive.
* Participant has clear ocular media and adequate pupillary dilatation in both eyes to allow for all imaging procedures, including good quality stereoscopic fundus photography and FAF.
* Participant has intraocular pressure (IOP) of ≤ 21 mmHg or less.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a women of childbearing potential (WOCBP).
  * WOCBP who has a negative serum pregnancy test at screening with a medical interview and agrees to follow the contraceptive guidance from the time of informed consent through at least 40 days after final study intervention administration.
* Female participant must not be breastfeeding or lactating starting at screening and throughout the investigational period and for 40 days after final study intervention administration.
* Female participant must not donate ova starting at first administration of study intervention and throughout the investigational period and for 40 days after final study intervention administration.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 40 days after final study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 40 days after final study intervention administration.
* Male participant must not donate sperm during the treatment period and for 40 days after final study intervention administration.
* Participant has ability to return for all study visits for the 12-month duration of the study.
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has evidence of choroidal neovascularization (CNV) in either eye.
* Participant has GA secondary to any condition other than AMD in the study eye (e.g., drug-induced).
* Participant has any ocular condition in the study eye that would progress during the course of the study and that could affect central vision or otherwise be a confounding factor.
* Participant has the presence of intraocular inflammation (≥ trace cell or flare), macular hole, pathologic myopia, epiretinal membrane, evidence of significant vitreomacular traction, vitreous hemorrhage or aphakia (pseudophakia with or without an intact capsule is not an exclusion criteria) in the study eye.
* Participant has the presence or history of idiopathic or autoimmune-associated uveitis in either eye.
* Participant has significant media opacities, including cataract, which might interfere with visual acuity (VA), assessment of toxicity or retinal imaging (fundus photography, FAF, spectral domain optical coherence tomography [SD-OCT], enhanced depth imaging optical coherence tomography [EDI OCT], fluorescein angiography [FA] or indocyanine green angiography [ICGA]) in the course of the study in either eye. Participant should not be entered if there is likelihood that they will require cataract surgery in either eye during the study.
* Participant has the presence of other causes of CNV, including pathologic myopia, high myopia (spherical equivalent of -8 diopters or more, or axial length of 25 mm or more), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, and multifocal choroiditis in either eye.
* Participant has any ocular or periocular infection (including blepharitis), or ocular surface inflammation in past 12 weeks in the study eye.
* Participant has any sign of diabetic retinopathy in either eye.
* Participant has BCVA of 20/320 or worse in the fellow eye.
* Participant has any prior treatment for AMD (dry or wet) or any prior intravitreal (IVT) treatment for any indication in either eye, except oral supplements of vitamins and minerals.
* Participant has concomitant treatment with any ocular or systemic medication that is known to be toxic to the lens, retina, or optic nerve in either eye (including, but not limited to amiodarone, deferoxamine, chloroquine/hydroxychloroquine sulfate, tamoxifen, phenothiazines, ethambutol or fingolimod).
* Participant has had any intraocular surgery or thermal laser treatment in the study eye within 3 months prior to screening, or any prior thermal laser treatment in the macular region, regardless of indication in the study eye.
* Participant has a history of any of the following procedures in the study eye: posterior vitrectomy, filtering surgery (e.g. trabeculectomy), glaucoma drainage device, corneal transplant, or retinal detachment.
* Participant has any previous therapeutic radiation in the region of the study eye.
* Participant has a present or previous history of participation in a study of ASP3021.
* Participant has a history of systemic treatment with any anti-complement agent in past or the likelihood of treatment with any systemic anti-complement agent during the study.
* Participant has received any investigational therapy within 60 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has a history or evidence of severe cardiac disease (e.g., New York Heart Association [NYHA] Functional Class III or IV, or history or clinical evidence of unstable angina, acute coronary syndrome, myocardial infarction or revascularization within last 6 months, or ventricular tachyarrhythmias requiring ongoing treatment.
* Participant has a history or evidence of clinically significant peripheral vascular disease, such as intermittent claudication or prior amputation.
* Participant has clinically significant impaired renal (serum creatinine > 2.5 mg/dL or status post-renal transplant or receiving dialysis) or hepatic function. Participants with these conditions may be enrolled after consultation with the medical monitor.
* Participant has a history of stroke within 12 months prior to screening.
* Participant has had any major surgical procedure within 1 month prior to screening.
* Participant has any condition that makes the participant unsuitable for study participation.
* Participant has a known or suspected serious allergy to the fluorescein dye and/or the indocyanine green dye used in angiography, povidone-iodine or hypersensitivity to ASP3021 or any components of the formulation used.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | Up to 12 Months
  An Adverse Event (AE) is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
  TEAEs are defined as an AE observed after first administration of ASP3021 until 30 days after final administration of ASP3021.
Number of participants with Serious TEAEs | Up to 12 Months
  A Serious Adverse Event is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other situations.
  TEAEs are defined as an AE observed after first administration of ASP3021 until 30 days after final administration of ASP3021.

SECONDARY OUTCOMES:
Number of participants with intraocular pressure (IOP) abnormalities and/or AEs | Up to 12 months
  Number of participants with potentially clinically significant IOP values.
Number of participants with ophthalmic examination abnormalities and/or AEs | Up to 12 months
  Number of participants with potentially clinically significant ophthalmic examination values.
Number of participants with laboratory value abnormalities and/or AEs | Up to 12 months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital signs abnormalities and/or AEs | Up to 12 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with 12-lead electrocardiogram (ECG) abnormalities and/or AEs | Up to 12 months
  Number of participants with potentially clinically significant 12-Lead ECG values.
Mean rate of growth (slope) over 12 months | Up to 12 months
  The growth (slope) over 12 months is estimated based on Geographic Atrophy (GA) area measured by fundus autofluorescence (FAF) (square root transformation).
Change from baseline in best corrected visual acuity (BCVA) | Baseline and up to 12 months
  BCVA will be measured by Early Treatment Diabetic Retinopathy Study [ETDRS] letters chart.
Change from baseline in low luminance best corrected visual acuity (LL BCVA) | Baseline and up to 12 months
  LL BCVA will be measured by ETDRS letters chart.
Number of participants with antidrug antibodies (ADA) status | Up to 12 months
  ADA will be recorded from the serum samples collected.
Number of participants with neutralizing antibodies (NAb) status for participant with positive ADA | Up to 12 months
  NAb will be recorded from the serum samples collected.
PK of ASP3021 in plasma: Concentration | Up to 2 months
  Concentration will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of ASP3021 in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to 12 months
  Ctrough will be recorded from the pharmacokinetic (PK) plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Inc
Locations (15):
- Japan (15):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - University of the Ryukyus hospital, Ginowan-shi, Okinawa
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - The University of Osaka Hospital, Suita-shi, Osaka
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Nihon University Hospital, Chiyoda-ku, Tokyo
  - Toyama University Hospital, Toyama, Toyama
  - University Of Yamanashi Hospital, Chuo-shi, Yamanashi

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.